CLINICAL TRIAL: NCT07009483
Title: Effectiveness of Psychodermatologic Educational Modules on Atopic Dermatitis Patient Outcomes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00153557
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Atopic Dermatitis (AD)
Keywords: Atopic Dermatitis; Dermatology; Psychodermatology; Patient Education
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational Module Arm (Experimental): This arm consists of participants living with atopic dermatitis that will be trialing our educational modules. In addition to receiving standard medical care, they will be asked to complete these modules throughout the duration of the study period.
  Interventions: Behavioral: Patient education modules providing information on the psychological aspects of atopic dermatitis treatment and management.
- Control Arm (No Intervention): This arm will consist of participants living with atopic dermatitis. They will receive standard medical care, but will not be given access to the educational modules until the study period has been completed.

INTERVENTIONS:
Behavioral: Patient education modules providing information on the psychological aspects of atopic dermatitis treatment and management. — Provision of online patient educational modules (in addition to patients receiving regular clinical action/ appointments at the Kaye Edmonton Clinic, the Stollery Children's Hospital, and the Rao Dermatology Clinic for Atopic Dermatitis).
  Arms: Educational Module Arm

SUMMARY:
In a previous part of this study, we created educational modules about the psychodermatology of inflammatory skin conditions, with a particular emphasis on atopic dermatitis, for patients. These modules will empower patients to better manage both the psychological and physical aspects of their skin conditions. As part of this project, we aim to conduct a clinical trial to determine the effectiveness of these modules on eczema severity and health-related quality of life in patients. We hope to use these findings to develop and disseminate accessible educational material on the psychological aspects of dermatologic care.

ELIGIBILITY:
Inclusion Criteria:

1. New diagnosis or follow-up for previous diagnosis of Atopic Dermatitis.
2. Reliable internet access to be able to access the e-modules.
3. Able to speak English at a level required to understand the content of this study.
4. Child participants will be included in this study contingent on the consent of their guardian/caregiver(s).
5. Age range of eligible participants: Age 4 years and older.

Exclusion Criteria:

1. Does not have a new diagnosis or follow-up for previous diagnosis of Atopic Dermatitis.
2. Unable to access and/or navigate e-modules with reasonable support/instruction.
3. Unable to speak English at a level required to understand the content of this study.
4. Unable to provide informed consent.
5. Less than 4 years of age.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Health-Related Quality of Life | Baseline, 4 weeks, and 12 weeks
  Quality of Life will be measured using the Dermatology Life Quality Index (DLQI). The scores range from 0 to 30 (higher score indicative of worse outcomes)

SECONDARY OUTCOMES:
Eczema Disease Severity | Baseline, 4 weeks, and 12 weeks
  Eczema Disease Severity will be measures using the Patient-Oriented SCORing for Atopic Dermatitis (PO-SCORAD). Scores range between 0 and 103 points (higher score indicative of worse outcomes)

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Dytoc, MD, PhD, FRCPC, Principal Investigator — University of Alberta
Locations (3):
- Canada (3):
  - Rao Dermatology, Edmonton, Alberta
  - Kaye Edmonton Clinic, Edmonton, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No
Not necessary

REFERENCES:
- [Background] Liu C, Chan M, Beard V, Mathura P, Dytoc M. Beyond Skin Deep: case-based online modules to teach multidisciplinary care in dermatology among clerkship students. BMC Med Educ. 2023 Feb 4;23(1):90. doi: 10.1186/s12909-023-04072-z. PMID 36739386
- [Background] Verma L, Turk T, Dennett L, Dytoc M. Teledermatology in Atopic Dermatitis: A Systematic Review. J Cutan Med Surg. 2024 Mar-Apr;28(2):153-157. doi: 10.1177/12034754231223694. Epub 2024 Jan 11. PMID 38205736
- [Background] Odeshi O, Turk T, Fiorillo L, Lowe S, Dytoc M. Teledermatology Versus In-Person Visits for the Follow-Up of Atopic Dermatitis Patients. J Cutan Med Surg. 2024 Jul-Aug;28(4):346-351. doi: 10.1177/12034754241253192. Epub 2024 May 28. PMID 38807447
- [Background] Turk T, Fujiwara E, Abba-Aji A, Mathura P, Dytoc M. Psychodermatology in Canada: A National Survey Assessment of Dermatologists' Perception, Practice Patterns, and Challenges. J Cutan Med Surg. 2021 May-Jun;25(3):249-256. doi: 10.1177/1203475420977473. Epub 2020 Dec 2. PMID 34039041
- [Background] Silverberg JI, Gelfand JM, Margolis DJ, Boguniewicz M, Fonacier L, Grayson MH, Ong PY, Chiesa Fuxench ZC, Simpson EL. Symptoms and diagnosis of anxiety and depression in atopic dermatitis in U.S. adults. Br J Dermatol. 2019 Sep;181(3):554-565. doi: 10.1111/bjd.17683. Epub 2019 Mar 5. PMID 30838645
- [Background] Silverberg JI, Gelfand JM, Margolis DJ, Boguniewicz M, Fonacier L, Grayson MH, Simpson EL, Ong PY, Chiesa Fuxench ZC. Patient burden and quality of life in atopic dermatitis in US adults: A population-based cross-sectional study. Ann Allergy Asthma Immunol. 2018 Sep;121(3):340-347. doi: 10.1016/j.anai.2018.07.006. Epub 2018 Jul 16. PMID 30025911
- [Background] Dalgard FJ, Gieler U, Tomas-Aragones L, Lien L, Poot F, Jemec GBE, Misery L, Szabo C, Linder D, Sampogna F, Evers AWM, Halvorsen JA, Balieva F, Szepietowski J, Romanov D, Marron SE, Altunay IK, Finlay AY, Salek SS, Kupfer J. The psychological burden of skin diseases: a cross-sectional multicenter study among dermatological out-patients in 13 European countries. J Invest Dermatol. 2015 Apr;135(4):984-991. doi: 10.1038/jid.2014.530. Epub 2014 Dec 18. PMID 25521458